CLINICAL TRIAL: NCT00701311
Title: An Open-Label Study of CC-10004 for Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-135
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Prostatitis; Chronic Prostatitis With Chronic Pelvic Pain Syndrome
Keywords: Prostatitis; Pelvic pain
MeSH Terms: conditions — Prostatitis; Pelvic Pain | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Drug CC-10004 (Experimental): Study drug CC-10004 20mg taken orally twice a day.
  Interventions: Drug: CC-10004

INTERVENTIONS:
Drug: CC-10004 — CC-10004 20 mg per day

SUMMARY:
Prostatitis is the most common urologic diagnosis in men under the age of 50 and the third most common diagnosis in older men. In Chronic Prostatitis (CP) or Chronic Pelvic Pain Syndrome (CPPS), men have lower urinary tract symptoms, pelvic pain, sexual dysfunction and decreased quality of life. Little is known about the cause of CP/CPPS. Likewise, no definitive therapy exists for CP/CPPS. We plan to study the use of CC-10004 in men with CP/CPPS.

DETAILED DESCRIPTION:
Prostatitis is the most common urologic diagnosis in men under the age of 50 and the third most common diagnosis in older men. In Chronic Prostatitis (CP) or Chronic Pelvic Pain Syndrome (CPPS), men have lower urinary tract symptoms, pelvic pain, sexual dysfunction and decreased quality of life.

Little is known about the cause of CP/CPPS. Likewise, no definitive therapy exists for CP/CPPS. Unlike bacterial prostatitis, where a clear infecting organism can be determined, CP/CPPS is not always treated with antibiotics.

Due to the significant inflammatory nature of CP/CPPS, most prior therapies have focused on targeting the inflammation. CC-10004 in several studies has shown to be an inhibitor of inflammatory mediators, and may decrease the pain experienced from CP/CPPS.

ELIGIBILITY:
Inclusion Criteria:

* Must be male aged ≥ 18 years at time of consent
* Must understand and voluntarily sign an informed consent form
* Male subjects with at least 3 months of symptoms of CP/CPPS (pain in the pelvic area, penis, scrotum, or perineum) who are refractory to other therapies (e.g. NSAIDS)
* Must be able to adhere to the study visit schedule and other protocol requirements
* Diagnosis of Chronic Prostatitis with a Chronic Prostatitis Symptom Index of at least 15/24
* Must meet the following laboratory criteria:

  * Hemoglobin > 9 g/dL
  * Hematocrit ≥ 27%
  * White blood cell (WBC) count ≥ 3000 /mL (≥ 3.0 X 109/L) and < 20,000/mL (< 20 X 109/L)
  * Platelets ≥ 100,000 /mL (≥ 100 X 109/L)
  * Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
  * Total bilirubin £ 2.0 mg/dL
  * Aspartate transaminase (AST) serum glutamic oxaloacetic transaminase (SGOT), and alanine transaminase (ALT) serum glutamate pyruvic transaminase,(SGPT), < 1.5x upper limit of normal (ULN)
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with female capable of becoming pregnant while on study medication and for 28 days after taking the last dose of study medication

Exclusion Criteria:

* Subjects who are female.
* Subjects with a documented positive urine culture within the past three months
* Subjects with duration of symptoms less than three months
* Subjects with genital infections within the past three months
* Subjects with clinical epididymitis within the past three months
* Subjects with known active or prior genitourinary cancers including renal, ureteral, bladder or prostate
* Subjects having received prior radiation to the abdominal or pelvic area
* Subjects with known bladder or ureteral calculi
* Subjects unable to complete a voiding diary
* Subjects with neutropenia (ANC < 750/ mm3)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study or confounds the ability to interpret data from the study
* History of active Mycobacterium tuberculosis infection (any subspecies) within 3 years prior to the screening visit. Infections that occurred > 3 years prior to entry must have been effectively treated.
* Positive Tuberculin skin test (Mantoux test)
* Clinically significant abnormality on the chest x-ray (CXR) at screening
* Any clinically significant abnormality on 12-lead ECG at screening
* Use of any investigational medication within 28 days prior to randomization or 5 half-lives if known (whichever is longer)
* History of malignancy within previous 5 years (except for treated basal-cell skin carcinoma(s) and/or fewer than 3 treated squamous-cell skin carcinomas)
* Subjects currently taking chemotherapeutic agents
* Positive human immunodeficiency virus (HIV), hepatitis B, or hepatitis C laboratory test result indicating active infection at screening.
* Subjects with known history of significant disease as determined by the PI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place over approximately one year from the offices of private urologists.
Pre-assignment Details: A total of 21 male subjects meeting inclusion criteria were recruited. Of these, two failed screening and two were enrolled but did not start drug. Therefore 17 subjects started treatment drug.
Groups:
- CC-10004: CC-10004 administered 20mg po twice daily for up to 12 weeks.
Period: Overall Study
Arm/Group | CC-10004
Started | 17
Completed | 9 (Eight subjects did not complete full period of treatment but their data was included in analysis.)
Not Completed | 8
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | CC-10004
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Global Response Assessment
Description: The primary efficacy measure was a Global Response Assessment (GRA), a subject completed questionnaire that measures improvement in overall symptoms on a 7-point scale: Markedly Improved - 7, Moderately Improved - 6, Mildly Improved - 5, Same - 4, Mildly Worse - 3, Moderately Worse - 2, Markedly Worse - 1.
  The primary outcome showing response to treatment was the number of subjects that were moderately or markedly improved on the GRA scale.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | CC-10004
Number analyzed (Participants) | 17
participants | 2

ADVERSE EVENTS:
Groups:
- Treatment Arm: Open label, one arm study.
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 12/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=17)
Nausea (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Facial Flushing (Vascular disorders) | 1
Lower extremity ulcer (Skin and subcutaneous tissue disorders) | 1
Mouth Ulcer (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The limitation of this study is that only 9 of 17 participants completed full 12 weeks of treatment and there was no placebo arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes